CLINICAL TRIAL: NCT02201537
Title: Non-invasive Diagnosis of Chronic Kidney Disease in Renal Transplants Kidney Transplanted Using Ultrasound Functional Imaging
Brief Title: Kidney Disease and Ultrasound Imaging
Acronym: Imag-NCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation de l'Avenir (Other); Bracco Imaging S.p.A. (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2012-A01070-43
Record Dates: First submitted 2014-07-17; First posted 2014-07-28 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Recipient of Kidney Transplant
Keywords: Ultrasound functional imaging; Chronic kidney Nephropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imag-NCT (Other): The ultrasound functional imaging will be performed at J15 (before the patient is discharged from service Transplantation) and at 3 and 12 months after the transplant.
  The functional imaging examinations will be held as follows:
  * 1st stage - the conventional Doppler ultrasound:
  * 2nd stage - the elastography:.
  * Step 3 - CEUS: It is performed on an ultrasound machine with a specific module with the same probes as conventional ultrasound. It requires the injection of 1.5 ml of SonoVue ®, a contrast ultrasound.
  Renal biopsy will be performed after the functional ultrasound at 3 and 12 months.
  Interventions: Device: renal echography

INTERVENTIONS:
Device: renal echography — Renal biopsy will be performed at 3 and 12 months.
  The functional imaging examinations will be held as follows:
  Step 1: the conventional Doppler ultrasound Step 2: ultrasound elastography Step 3: CEUS

SUMMARY:
The hypothesis of our study is that a correlation exists between the couple ultrasound elastography- renal perfusion estimated with contrast-enhanced ultrasound and the degree of fibrosis estimated in a semi-quantitative way in 4 stages (0; 25 %; 25-50 %; > 50 %), as elastography alone did not allow to differentiate moderated fibrosis at 3 months in our feasibility study.

DETAILED DESCRIPTION:
Kidney transplant patients are exposed to long-term immunosuppressive therapy, and have an increased risk of infections and cancer, while a lack of treatment increases the risk of rejection. The development of imaging techniques to characterize the status of the graft remains a challenge in transplantation. Ideally, they should identify complications (acute rejection, chronic allograft nephropathy, nephrotoxicity ...) without the need for invasive procedures and thus lead to better customization of immunosuppressive therapy.

The post-transplant follow-up is based on the monitoring of graft function. Impaired function suggests the possibility of a complication, but requires confirmation by an invasive procedure such as renal biopsy. In addition, the diagnosis remains complex at a relatively advanced stage of the process due to damage to the graft parenchyma. To anticipate the altered function and detect subclinical lesions, screening biopsies have been used to diagnose chronic rejection. By definition, screening for subclinical lesions can not be based on any biological parameter; the diagnosis of subclinical complications thus requires performing multiple systematic biopsies, which are scheduled at 3 months and 1 year.

Doppler ultrasound is an imaging method of choice for the study of renal transplant, but it cannot diagnose the NCT due to the absence of specific findings. The lack of early diagnostic test for NCT is a major obstacle to the development and evaluation of new therapeutic options to prevent, slow or stabilize renal fibrosis. It is therefore necessary to develop a non-invasive imaging technique for the early diagnosis of NCT.

Ultrasound elastography is a technique that allows tissue stiffness measurements and provides a parametric picture.

The main objective of our study is to evaluate the performances of elastography and measurement of renal perfusion (area under the ROC curve) to diagnose the NCT and determine for each both measures a threshold to maximize the sensitivity. These performances will be evaluated at 3 months and 12 months. The results can also be compared to other imaging modalities such as functional MRI, and to clinical events (obstruction, infection…).

Functional ultrasound imaging should identify diagnostic and prognostic criteria of NCT, and enable the development of less invasive therapeutic protocols to evaluate new therapeutic approaches

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patient with informed consent;
* Recipient of a living donor graft or cadaveric donor patient;
* No contraindication for biopsy of the graft;
* No contraindication to the injection of SonoVue ®:

  * hypersensitivity to sulfur hexafluoride
  * acute coronary syndrome, unstable ischemic heart disease (myocardial infarction phase formation or evolution, typical resting angina in the previous 7 days, significant worsening of cardiac symptoms in the previous 7 days, recent intervention on the coronary arteries or another factor suggesting clinical instability (eg, recent deterioration of ECG changes in clinical or laboratory parameters), acute heart failure, stage III or IV heart failure, severe arrhythmias.
  * right-left shunt, severe pulmonary hypertension (PAP> 90 mmHg), uncontrolled systemic hypertension, respiratory distress syndrome
* Affiliated to a social security scheme

Exclusion Criteria:

* Refusal to participate in the study;
* Inability / refusal to give informed consent;
* contraindication for biopsy testing graft;
* Presence of a contraindication to the injection of SonoVue ®.
* Presence of a peripheral venous access in a non-restricted already infused patient, not pickable under ultrasound
* Breastfeeding, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2013-03-19 (Actual); Primary Completion 2016-03-19 (Actual); Study Completion 2016-03-19 (Actual)

PRIMARY OUTCOMES:
renal Elastography | 3 months
  The assessment of renal function is performed by the serum creatinine and calculation of glomerular filtration rate estimated by the formula Modified Diet in Renal Disease (MDRD) 4-parameter at 3 and 12 months post-transplantation. In addition, a measure of glomerular filtration rate using the technique to iohexol is performed routinely at 12 months post-transplant as part of routine monitoring of transplant patient.
  The ultrasound functional imaging will be performed at 15 days, 3 and 12 months after transplantation.
  The functional imaging examinations will be held as follows:
  Step 1: the conventional Doppler ultrasound 2nd step: the ultrasound elastography Step 3 : CEUS
Renal Elastography and contrast-enhanced US | 12 months
  The assessment of renal function is performed by the serum creatinine and calculation of glomerular filtration rate estimated by the formula Modified Diet in Renal Disease (MDRD) 4-parameter at 3 and 12 months post-transplantation. In addition, a measure of glomerular filtration rate using the technique to iohexol is performed routinely at 12 months post-transplant as part of routine monitoring of transplant patient.
  The ultrasound functional imaging will be performed at 15 days, 3 and 12 months after transplantation.
  The functional imaging examinations will be held as follows:
  Step 1: the conventional Doppler ultrasound 2nd step: the ultrasound elastography Step 3 : CEUS

SECONDARY OUTCOMES:
renal Elastography | 3 months
  Correlation between elastography and renal function with degree of fibrosis and renal function will be calculate using Pearson coefficient of correlation
Correlation between renal elastography and perfusion and degree of fibrosis and renal function | 12 months
  Correlation between elastography and renal function with degree of fibrosis and renal function will be calculate using Pearson coefficient of correlation
renal Elastography in patients with chronic kidney disease | 12 months
  this two measures will be express in evolution percentage at J15 and 3 months. The evolution percentage will be compared with imaging of patient with chronic kidney disease to determine if elastography and renal perfusion can predict chronic kidney disease at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel CORREAS, PUPH, Principal Investigator — Necker Hospital
Locations (1):
- NECKER Hospital, Paris, France